CLINICAL TRIAL: NCT07325474
Title: Development & Implementation of Culturally Sensitive Safety Planning to Reduce Suicide Risk in Adolescents Seeking Care in Rural Emergency Departments
Brief Title: Plan and Protect: Safety Planning for Teens in Rural Emergency Departments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, JoAnna K. Leyenaar, Professor of Pediatrics, Professor of the Dartmouth Institute, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02002568; 5R01NR021638-02 (NIH)
Record Dates: First submitted 2025-12-19; First posted 2026-01-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Suicide Ideation; Suicide Attempt
Keywords: Suicide; Safety Planning; Adolescent; Mental Health Services; Emergency Services
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Intervention Model Description: Stepped wedge randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plan & Protect (Experimental): Plan and Protect is a tablet-based program that integrates a youth-facing safety-planning module with a caregiver-facing home safety planning decision aid to create culturally sensitive, locally tailored safety plans and promote caregiver engagement in home safety during rural ED visits for adolescent suicidality
  Interventions: Behavioral: Plan & Protect safety planning intervention
- Care as usual (Other): Outcomes for adolescents and their caregivers enrolled during the pre-implementation (usual care) periods at each hospital will be compared to outcomes for those enrolled after their hospital implements the P&P program as quality improvement
  Interventions: Behavioral: Care as usual

INTERVENTIONS:
Behavioral: Plan & Protect safety planning intervention — Plan and Protect (P&P) is a tablet-based, family-centered quality improvement program targeted to rural Northern New England that combines a youth-facing safety-planning module with a caregiver-facing home safety decision aid and youth safety information. The goal is to help adolescents and their caregivers develop concrete, culturally-sensitive safety plans during emergency department visits.
  Arms: Plan & Protect
Behavioral: Care as usual — Adolescents and caregivers will receive treatment as usual at the Emergency Department.
  Arms: Care as usual

SUMMARY:
The goal of this observational study is to determine whether implementing a culturally sensitive, tablet-based safety planning program called Plan & Protect (P&P) within rural emergency departments can improve home safety and reduce suicide risk in adolescents presenting with suicidality.

The main questions it aims to answer are:

* Will implementing P&P increase caregiver-reported home safety (reduce access to firearms and unsafe medication storage) for adolescents 12-17 years old presenting to rural EDs with suicidal ideation, self-harm, or mental health crisis?
* Will implementing P&P decrease adolescent-reported perceived suicide risk and related outcomes (e.g., suicide events, and attendance at follow-up mental healthcare)?

Researchers will compare outcomes for adolescents and caregivers receiving P&P (implemented as the new standard of care at sites during the intervention periods) to those receiving usual care (prior to P&P implementation at those hospitals) to see if P&P increases home safety and decreases suicide risk and related healthcare utilization.

Participants will, if clinically appropriate:

* Complete the tablet-based P&P modules during their ED visit
* Complete self-report measures at baseline, ~30 days, and ~3 months post-discharge
* A subset will also participate in semi-structured interviews

DETAILED DESCRIPTION:
One-in-five children and adolescents in the United States (US) live in rural areas where they are more likely to live in poverty, have neurodevelopmental, behavioral and mental health conditions, and die during childhood than their urban-residing peers. Suicide is a leading cause of childhood mortality, and rural-residing youth are two times more likely to die from suicide than urban-residing youth. Nearly half of children and adolescents with mental health conditions do not receive treatment, and those in rural areas face unique barriers to care due to geographic isolation, stigma, and shortages of pediatric services and clinicians. Given barriers to community-based mental healthcare, youth with suicidal ideation and/or suicide attempt (hereafter "suicidality") increasingly present to emergency departments (EDs) for care. However, most clinicians practicing in rural EDs are under-prepared and under-resourced to care for this population.

In order to fill this gap, this project aims to improve home safety and decrease suicide risk in youth 12-17 years of age who present to rural EDs with suicidal ideation or attempt, leveraging community-based participatory research approaches and technology to implement, with high fidelity, culturally-sensitive and nationally recommended safety planning procedures. To achieve this goal, we will integrate P&P, a culturally sensitive, tablet-based safety planning program as a quality improvement intervention at 4 hospitals in the Dartmouth Health network using a hospital-randomized stepped wedge design and will evaluate the program using a type 1 hybrid implementation-effectiveness design.

Aim: To determine the effectiveness of P&P compared to usual care for youth with suicidality and their caregivers to increase home safety and decrease suicide risk; evaluate the extent to which these outcomes are mediated by caregiver and youth self-efficacy and expectations of suicide risk; and assess the reach, effectiveness, adoption, implementation and maintenance of P&P using a mixed methods approach.

ELIGIBILITY:
Inclusion criteria for children:

* 12-17 years of age (and their parent/caregiver(s))
* Ability to speak and complete surveys in English
* History of emergency department visit for suicidality, self-harm or mental health crisis
* Medically stable

Exclusion criteria for children:

* Cognitive or developmental delays that preclude program participation based on clinical team assessment
* Diagnosis of psychosis
* Primary diagnosis of an eating disorder
* Parent/guardian not able to provide consent in English
* Clinical team concern for patient or staff safety based upon active behavioral concerns
* Parent/guardian not available to provide consent (e.g youth is in child protective custody/ward of the state)

Inclusion criteria for parents/caregivers:

* Parent or caregiver of an eligible child
* 18 years old or older
* Ability to speak and complete surveys in English

Exclusion criteria for parents/caregivers:

-Inability to understand key aspects of the study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 550 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Improved home safety (parent and youth) | 30 and 90 days after ED visit
  Reduced access to firearms and medications at home. This will be collected with five questions about presence of medications and firearms at home, if they are stored unlocked, and if firearms are loaded. We will measure improvement in safety across the time frame.
Concise Health Risk Tracking 9-item measure (youth) | 30 and 90 days after ED visit
  The Concise Health Risk Tracking (CHRT) is a 9-item survey that assesses suicidal thoughts and behaviors in the past week, with response options ranging 0-4. Total scores range 0-36, with higher scores indicating more severe suicidality.

SECONDARY OUTCOMES:
Suicide Events (youth) | 30 and 90 days after ED visit
  Four self-reported questions from the Youth Risk Behavior Survey focus on suicidal ideation, attempts, and attempt severity, augmented by electronic health record review for emergency room and hospital visits for suicide ideation and/or attempt and/or death.
Mental Health Care Utilization (parent and youth) | 30 and 90 days following ED visit
  Any mental or emotional health care received after their emergency department visit using a checklist adapted from nationally administered healthcare utilization surveys. Response categories (primary care, mental health provider, outpatient/urgent care, emergency department, school based care) were derived from health service use domains captured in the Medical Expenditure Panel Survey.
Reduced Access to Firearms at Home (parent and youth) | 30 and 90 days after ED visit
  Improved home safety with respect to firearm access. This will be collected with three questions about presence of firearms at home, if they are stored unlocked, and if they are loaded. We will measure improvement in safety across the time frame.
Reduced Access to Medications at Home (parent and youth) | 30 and 90 days after ED visit
  Improved home safety with safer storage of medications. This will be collected with two questions about presence of medications at home and if they are stored unlocked. We will measure improvement in safety across the time frame.

OTHER OUTCOMES:
Change in Parental Self-Efficacy to Support Teens During a Suicidal Crisis (parent) | 30 and 90 days after ED visit
  This 9-item scale measures parent confidence regarding their ability to engage in activities to prevent or assist their child in managing a suicidal crisis. Answer choices range from 0 (not at all confident) to 10 (completely confident), with an anchor of 5 (somewhat confident).
Change in Parental Perceptions of Teen Suicide Risk (parent) | 30 and 90 days after ED visit
  This 3-item measure looks at parental understanding of their teen's suicide risk. Answer choices range from 0 (not at all confident) to 10 (completely confident), with an anchor of 5 (somewhat confident).
Change in Patient Perceptions of Their Own Suicide Risk (youth) | 30 and 90 days after ED visit
  This 3-item self-report measure examines how at risk a patient believes they are. It is scored on a 5-point Likert from 0-4 where higher = greater perceived risk and has a total possible score of 15.
Change in Efficacy to Cope with Suicidal Thoughts and Urges Scale (youth) | 30 and 90 days after ED visit
  The Efficacy to Cope with Suicidal Thoughts and Urges Scale was designed to measure children's abilities to manage suicide-related thoughts and impulses. It contains 10 coping skills and children rate their confidence in their ability to use each coping skill to manage their suicidality. Responses range from 0 to 10 with 0 = Not at all confident, 5 = Somewhat confident, and 10 = Extremely confident.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnna K Leyenaar, MD, PhD, MPH, Principal Investigator — Dartmouth College
Locations (4):
- United States (4):
  - Cheshire Medical Center, Keene, New Hampshire
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Alice Peck Day Memorial Hospital, Lebanon, New Hampshire
  - New London Hospital, New London, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded into the NIMH Data Archive (NDA).
  Data will be collected from approximately 275 adolescents 12-17 years of age and 275 parents or caregivers. Measures include:
  1. Sociodemographic characteristics of adolescents and caregivers
  2. Follow-up mental health care
  3. DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure for Youth Self-report
  4. Efficacy to Cope with Suicidal Thoughts and Urges Scale for Youth Self-report
  5. Self-Assessed Expectations of Suicide Risk for Youth
  6. Parental Self-Efficacy to Support Teens During a Suicidal Crisis
  7. Concise Health Risk Tracking - Self-Report (CHRT-SR)
  8. Caregiver and adolescent-reported firearms in home/on property (yes/no) and firearm storage practices
  9. Caregiver- and adolescent-reported medications in home (yes/no) and medication storage practices
Supporting Information: Study Protocol
Time Frame: All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: Per NDA access requirements and protocols.